CLINICAL TRIAL: NCT06484283
Title: Investigation of the Effect of Meditation Applied to Mothers With Oncology-Diagnosed Children on Mothers' Resilience and Spiritual Well-Being Levels: A Randomized Controlled Study
Brief Title: The Effect of Meditation on Resilience and Spiritual Well-Being Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Eda Simsek Sahin, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-45778635-050.99-144574
Record Dates: First submitted 2024-06-07; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Well-Being, Psychological
Keywords: Oncology; Meditation; Resilience; Spiritual Well-Being
MeSH Terms: conditions — Psychological Well-Being; Neoplasms | interventions — Meditation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Researchers will inform mothers who apply to the unit and invite them to participate in the study. The informed consent form will be read to mothers who accept the study, and their written consent will be obtained. A simple randomization method will be used to control selection bias that may arise while determining research groups. All study participants (intervention and control groups) will be asked to complete the Introductory Characteristics Form, Spiritual Well-Being Scale, and Connor Davidson Resilience Scale Short Form. After this stage, mothers in the intervention group will be given a meditation application video, and the details of the application (how long and how to meditate) will be explained. After the implementation period, the mothers will be again administered the Spiritual Well-Being Scale and the Connor Davidson Resilience Scale Short Form
  Interventions: Other: Meditation
- Control Group (No Intervention): No intervention will be made to the control group. To act ethically, after data is collected from the experimental and control groups, participants in the control group will be given the meditation video to practice.

INTERVENTIONS:
Other: Meditation — Guided meditation will be applied within the scope of the study. A guided meditation video prepared by a Yoga Alliance-certified researcher will be used for this intervention. Guided meditation aims to ensure being in the moment (here and now) with the help of breathing. Meditation practice will take participants 10 minutes.
  Arms: Experimental Group

SUMMARY:
Childhood cancers have become an important health problem with a rapidly increasing incidence. Although global and national data show that the developmental status of countries has an impact on the success of treatment, there is a significant increase in the incidence of childhood cancers. With the diagnosis of childhood cancer, long-term and exhausting treatments, increased financial and moral burdens and psycho-social difficulties affect children, but it is inevitable that the child's parents are also affected by the situation. Childhood cancer has serious effects on the physical and psychological health of pediatric patients, their families and caregivers. In this process, parents may face psychosocial problems such as depression, anxiety, stress, fatigue, burnout, disruption of family dynamics and inadequacy. Although the treatment process affects the adaptation, coping and family dynamics of all family members, it can be much more tiring and exhausting for mothers, who are often the primary caregivers of the child.Studies point out that parents of a child with oncology need to adapt to the long and strenuous treatment procedures in order to cope and cope with these challenges. Adaptation involves parents more quickly in integrating and taking an active role in the treatment and care processes. This has been linked to people's ability to be resilient. Although resilience is an ability that develops over time, it is very important to support the family of parents of children diagnosed with oncology in this sense. Meditation is a practice with ancient teachings dating back at least 3000 years. In recent years there has been a growing interest in its benefits for psychological and spiritual well-being in many fields including medicine, nursing, psychology, sociology and education. Although it has a wide variety of definitions and contents, it generally consists of practices such as attention and focus training for mindfulness, breathing and relaxation practices for relaxation, and attention practices for mental calming. Studies show that meditation practices are used for purposes such as individual and psychological well-being, anxiety, depression, strengthening spirituality and positive results are obtained. This study aims to determine the effects of meditation on the spiritual well-being and resilience levels of mothers with oncologically diagnosed children aged 6-18 years.

DETAILED DESCRIPTION:
Meditation is a practice that dates back at least 3000 years and has ancient teachings. In recent years, there has been increasing interest in its benefits for psychological and spiritual well-being in many fields, including medicine, nursing, psychology, sociology, and education. Although it has various definitions and contents, it generally consists of practices such as attention and focus training for awareness, breathing and relaxation practices for relaxation, and attention practices for mental calming. Studies show that meditation practices are used for purposes such as individual and psychological well-being, anxiety, depression, and strengthening spirituality, and positive results are obtained. It is the responsibility of nurses to protect and support parents from distressing and tiring processes such as having a child diagnosed with oncology, caring for the child, and interrupting family processes. Nurses are among the most active participants in the process, working with parents and the child throughout the entire process, starting from the child's diagnosis. Examining and evaluating parents' spiritual strength and resilience and intervening in time is very important. This research was planned to investigate the spiritual well-being and resilience of mothers with children diagnosed with oncology and to determine and evaluate the effect of meditation practice on these parameters. So, what can we do to empower parents of children diagnosed with oncology? Plans to contribute to the literature on the subject. Contributing to a particular field, such as pediatric oncology, will support nurses working in these units to develop a more comprehensive and holistic approach and improve their quality of care. Quality care will positively support, strengthen and guide the child and the parents on this journey.

ELIGIBILITY:
Inclusion Criteria:

* Mothers whose children have been diagnosed with oncology,
* Mothers whose children have received at least one course of chemotherapy
* Mothers who can speak and understand Turkish
* Mothers who volunteer to participate in the study will be included.

Exclusion Criteria:

* Mothers who have a particular problem that prevents communication (neurodevelopmental delay, verbal speech difficulty, hearing or hearing problems),
* Mothers who are being treated for relapse or whose children are in the terminal stage will be excluded from the study.

Ages: 6 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Women in the 6-18 age group with children diagnosed with oncology will be included in the study.
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Spiritual well-being level (measured by "Spiritual Well-being Scale".It is a five-point Likert scale comprising 29 items in three sub-dimensions. The score that can be obtained from the scale varies between 29 and 145.) | Measurements will be taken at registration, when participants are included in the study, and 3 weeks after the first measurement.
  The effect of meditation applied to mothers with children with oncological diagnosis in the 6-18 age group on their spiritual well-being level.
Resilience level (measured by the Connor Davidson Resilience Scale Short Form. The scores that can be obtained from the scale vary between 0 and 40. High scores obtained from the scale are considered as high psychological resilience.) | Measurements will be taken at registration, when participants are included in the study, and 3 weeks after the first measurement.
  The effect of meditation applied to mothers with children with oncological diagnosis in the 6-18 age group on their resilience level.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, İ̇zmi̇t, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans to roll out IPD.